CLINICAL TRIAL: NCT07273188
Title: Gallium-68-labeled Fibroblast Activation Protein Inhibitor-46 (68Ga-FAPI-46) PET in Crohn's Disease Patients: a Case-control Study Designed to Illuminate the Spectrum of Fibrostenosis in Patients With Small Bowel Crohn's Disease
Brief Title: 68Ga-FAPI-46 PET/CT for Assessing Small Bowel Fibrostenosis in Crohn's Disease
Acronym: FAPI-PETCD
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other)
Responsible Party: Principal Investigator, David J. Bartlett, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 25-008885
Record Dates: First submitted 2025-11-24; First posted 2025-12-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Crohn's Disease; Intestinal Fibrosis; Inflamatory Bowel Disease; Intestinal Strictures Related to Crohn´s Disease
Keywords: Ga68-FAPI-46; PET/CT; Small bowel stricture; Fibrostenosis; FAPI PET; Small bowel Crohn's disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- A group of participants getting PET/CT scan with 68Ga-FAPI-46 (Experimental): Ga68-FAPI-46 radioactive tracer binding to FAP
  Interventions: Drug: Ga68-FAPI-46

INTERVENTIONS:
Drug: Ga68-FAPI-46 — Gallium-68-labeled fibroblast activation protein inhibitor-46 (68Ga-FAPI-46) , 5 mCi ±10%, IV

SUMMARY:
This study is a prospective, case-control study evaluating whether the PET radiotracer 68Ga-FAPI-46 can detect fibrostenosing Crohn's disease in the small bowel. The goal is to determine whether areas of early or developing fibrosis ("pre-stricture" changes) demonstrate uptake of the tracer, which binds to fibroblast activation protein (FAP).

Participants with small bowel Crohn's disease will be assigned to either a case or control group based on CT or MR enterography findings at enrollment.

Cases will include participants who have a small bowel stricture or probable stricture, with or without penetrating complications.

Controls will include participants with small bowel Crohn's disease without strictures. Controls may have active inflammatory disease, luminal narrowing, or no active inflammation (including postoperative or chronic changes), as long as no stricture is present.

Because most radiologic strictures represent more advanced fibrostenosis, the study aims to enroll a larger proportion of controls to better characterize early fibrotic changes. Approximately one-third to one-half of participants will be cases, and the remainder controls. This design will allow comparison of FAPI uptake patterns in patients with and without strictures to understand how FAP expression relates to the development of small bowel fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Known small bowel Crohn's disease
* Research or clinical MR enterography, or clinical CT enterography, within 3 months.
* Male or female with age greater than 18 years old.
* Diagnosis of Crohn's disease by a gastroenterologist
* Willingness to undergo 68Ga-FAPI-46 PET/CT
* Subjects with the capacity to give informed consent and willingness to provide written consent

Exclusion Criteria:

* Pregnant and/or breast-feeding subjects.
* Hypersensitivity to any excipients in 68Ga-FAPI-46

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-01-26 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Completion of PET/CT with Ga68-FAPI-46 by all participants | Through study completion, an average of 2 years
Number of participants completing PET/CT with Ga68-FAPI-46 | Through study completion, an average of 2 years
  Participants complete PET/CT with Ga68-FAPI-46

CONTACTS AND LOCATIONS:
Overall Officials: David J Bartlett, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No